CLINICAL TRIAL: NCT00987454
Title: A Randomised, Placebo-controlled Trial of Erythropoietin in ICU Patients With Traumatic Brain Injury
Brief Title: Erythropoietin in Traumatic Brain Injury (EPO-TBI)
Acronym: EPO-TBI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZIC-RC/RB002
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Epoetin Alfa; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Active Comparator): Epoetin alfa 40,000 international units will be given by subcutaneous injection to eligible patients, allocated to the treatment arm, on Study Days 1; 8 and15 during the intensive care unit stay.
  Interventions: Drug: Epoetin Alfa
- Placebo (Placebo Comparator): Sodium Chloride 0.9% in m/L will be given by subcutaneous injection to eligible patients, allocated to the placebo arm, on Study Days 1; 8 and15 during the intensive care unit stay.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Epoetin Alfa — 40,000 IU given as subcutaneous injection weekly up to 3 doses
  Other Names: Eprex
  Arms: Erythropoietin
Drug: Sodium Chloride 0.9% — 1 m/L given as subcutaneous injection weekly up to 3 doses
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This study seeks to determine if erythropoietin alpha (EPO) administered to adult critical care patients with moderate or severe traumatic brain injury improves neurological function assessed at six months after injury.

DETAILED DESCRIPTION:
Many people who have a traumatic brain injury (TBI) - usually from a blow to the head such as in a vehicle collision or in a fall do not survive or, if they do, suffer from long-term disability. Previous studies have shown that about 1,000 people in Australia and New Zealand suffer a moderate or severe TBI every year. With current best available treatment and therapies many of these patients sustain loss of brain function and long term disability in varying degrees.

When a patient sustains a traumatic brain injury there are two phases to the injury. First, the head-impact causes immediate damage to the brain. The secondary injury, which can evolve over hours or weeks, is a very complicated process. It involves many, linked, changes to the cells, brain chemistry, tissues or blood vessels that can destroy brain tissue. The treatment of brain injury focuses on trying to minimize the secondary injury and there is much research being done to try to find treatments that will prevent it.

Erythropoietin (EPO) has recently emerged as a drug that may help reduce secondary injury and improve brain function. It has been found to offer some protection to the brain when brain cells are deprived of their normal oxygen supply causing cells to die or be impaired.

The aim of this study is to determine if EPO reduces secondary brain injury and helps patients make a better recovery after traumatic brain injury. The investigators also plan to monitor the effect of EPO on the rate of deep vein thrombosis (DVT - blood clots in the large veins in lower extremity) in patients with moderate or severe TBI in the intensive care unit (ICU).

Study Hypothesis:

In patients with moderate (GCS 9-12) or severe (3-8) TBI, EPO therapy improves long-term neurological function assessed 6 months after injury.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 15 to ≤ 65 years of age
* Are < 24 hours since primary traumatic injury
* Are expected to stay ≥ 48 hours
* Have a haemoglobin not exceeding the upper limit of the applicable normal (ULN) reference range in clinical use at the treating institution
* Have written informed consent from legal surrogate

Exclusion Criteria:

* GCS = 3 and fixed dilated pupils
* History of DVT, PE or other thromboembolic event
* A chronic hypercoagulable disorder, including known malignancy
* Treatment with EPO in the last 30 days
* First dose of study drug unable to be given within 24 hours of primary injury
* Pregnancy or lactation or 3 months post partum
* Uncontrolled hypertension (systolic blood pressure of >200 mm Hg or diastolic blood pressure of >110 mm Hg)
* Acute myocardial infarct
* Expected to die imminently (< 24 hours)
* Inability to perform lower limb ultrasounds
* Known sensitivity to mammalian cell derived products
* Hypersensitivity to the active substance or to any of the additives
* Pure red cell aplasia (PRCA)
* End stage renal failure (receives chronic dialysis)
* Severe pre-existing physical or mental disability or severe co-morbidity that may interfere with the assessment of outcome
* Spinal cord injury
* Treatment with any investigational drug within 30 days before enrolment
* The treating physician believes it is not in the best interest of the patient to be randomised to this trial

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2010-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Combined proportion of unfavourable neurological outcomes at 6 months: severe disability (defined as GOSE scores 2-4) or death (GOSE score 1). | 6 months

SECONDARY OUTCOMES:
Probability of an equal or greater Glasgow Coma Scale Extended (GOSE) level at 6 months compared to the probability of a lesser GOSE level, using a proportional odds model | 6 months
Proportion of surviving patients with unfavourable neurological outcome (GOSE 2-4) at 6 months | 6 months
Quality of life assessment (SF-12 and EQ-5D) at 6 months | 6 months
Mortality at 6 months | 6 months
Rate of proximal deep venous thrombosis detected during screening by compression Doppler ultrasound | 21 days
Proportion of patients with composite thrombotic vascular events (DVT, pulmonary embolus, myocardial infarction, cardiac arrest and cerebrovascular events) at 6 months | 6 months
Cost effectiveness analysis at 6 months (based on EQ-5D) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alistair D Nichol, MD, Study Chair — Monash University
Locations (28):
- Australia (14):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - The Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hosptial, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- France (5):
  - Hôpital Michallon, Grenoble
  - Hôpital universitaire Caremeau, Nîmes
  - Hôpital Lariboisière, Paris
  - Hôpital de Bicêtre, Paris
  - CHU de Rouen, Rouen
- Johannes Gutenberg-Universtität, Mainz, Germany
- Beaumont Hospital, Dublin, Ireland
- New Zealand (4):
  - Auckland City Hospital, Auckland, North Island
  - Wellington Regional Hospital, Wellington, North Island
  - Christchurch Hospital, Christchurch, South Island
  - Dunedin Hospital, Dunedin
- King Fahad National Guard Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879
- [Derived] Skrifvars MB, Bailey M, Moore E, Martensson J, French C, Presneill J, Nichol A, Little L, Duranteau J, Huet O, Haddad S, Arabi YM, McArthur C, Cooper DJ, Bendel S, Bellomo R; Erythropoietin in Traumatic Brain Injury (EPO-TBI) Investigators and the Australian and New Zealand Intensive Care Society (ANZICS) Clinical Trials Group. A Post Hoc Analysis of Osmotherapy Use in the Erythropoietin in Traumatic Brain Injury Study-Associations With Acute Kidney Injury and Mortality. Crit Care Med. 2021 Apr 1;49(4):e394-e403. doi: 10.1097/CCM.0000000000004853. PMID 33566466
- [Derived] Skrifvars MB, Moore E, Martensson J, Bailey M, French C, Presneill J, Nichol A, Little L, Duranteau J, Huet O, Haddad S, Arabi Y, McArthur C, Cooper DJ, Bellomo R; EPO-TBI Investigators and the ANZICS Clinical Trials Group. Erythropoietin in traumatic brain injury associated acute kidney injury: A randomized controlled trial. Acta Anaesthesiol Scand. 2019 Feb;63(2):200-207. doi: 10.1111/aas.13244. Epub 2018 Aug 21. PMID 30132785
- [Derived] Nichol A, French C, Little L, Haddad S, Presneill J, Arabi Y, Bailey M, Cooper DJ, Duranteau J, Huet O, Mak A, McArthur C, Pettila V, Skrifvars M, Vallance S, Varma D, Wills J, Bellomo R; EPO-TBI Investigators; ANZICS Clinical Trials Group. Erythropoietin in traumatic brain injury (EPO-TBI): a double-blind randomised controlled trial. Lancet. 2015 Dec 19;386(10012):2499-506. doi: 10.1016/S0140-6736(15)00386-4. Epub 2015 Oct 6. PMID 26452709
- [Derived] Nichol A, French C, Little L, Presneill J, Cooper DJ, Haddad S, Duranteau J, Huet O, Skrifvars M, Arabi Y, Bellomo R; EPO-TBI Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Erythropoietin in traumatic brain injury: study protocol for a randomised controlled trial. Trials. 2015 Feb 8;16:39. doi: 10.1186/s13063-014-0528-6. PMID 25884605
- [Derived] Presneill J, Little L, Nichol A, French C, Cooper DJ, Haddad S, Duranteau J, Huet O, Skrifvars M, Arabi Y, Bellomo R; EPO-TBI Investigators; ANZICS Clinical Trials Group. Statistical analysis plan for the Erythropoietin in Traumatic Brain Injury trial: a randomised controlled trial of erythropoietin versus placebo in moderate and severe traumatic brain injury. Trials. 2014 Dec 20;15:501. doi: 10.1186/1745-6215-15-501. PMID 25528574
- [Derived] Moore EM, Bellomo R, Nichol AD. Erythropoietin as a novel brain and kidney protective agent. Anaesth Intensive Care. 2011 May;39(3):356-72. doi: 10.1177/0310057X1103900306. PMID 21675055